CLINICAL TRIAL: NCT06784128
Title: Impact of TECAR Therapy on Pain and Function in Adhesive Capsulitis: A Randomized Controlled Trial
Brief Title: Impact of TECAR Therapy on Pain and Function in Adhesive Capsulitis:
Acronym: TECAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Oznur Uzun, MD, Deputy Chief of Physical Medicine and Rehabilitation Hospital, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-3840; ANKARA BILKENT CITY HOSPITAL (Other: PHYSICAL MEDICINE AND REHABILITATION HOSPITAL)
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Pain Management; TECAR Therapy; VAS
MeSH Terms: conditions — Bursitis; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS combined with therapeutic exercise and hot pack (Control Group) (Active Comparator): TENS was employed as a non-invasive pain management technique in this study, utilizing the Intellect Advanced device manufactured by Chattanooga Group. Electrodes were strategically placed over the affected shoulder, ensuring coverage of the most painful areas as well as relevant nerve pathways to maximize the analgesic effect. A symmetric biphasic waveform was selected, with a frequency of 100 Hz and a pulse duration of 100 microseconds. The intensity of the stimulation was adjusted according to the patient's tolerance, typically aiming for a strong, yet comfortable tingling sensation.
  Interventions: Other: Therapeutic Exercise Program; Other: Hot Pack; Device: TENS
- TECAR combined with TENS and therapeutic exercise and hot pack (TECAR Group) (Experimental): In the experimental group, in addition to conventional TENS and hotpack, TECAR therapy was also applied three times per week for a total of six sessions. TECAR therapy was administered using the BTL-6000 TR-Therapy PRO device by an experienced physiotherapist.The device emitted energy at a frequency of approximately 500 kHz and used three types of electrodes: active, neutral, and static application electrodes. The active electrodes were of two types, capacitive and resistive, and were applied directly during treatment. The neutral electrode functioned as a reference and was positioned beneath the patient's body, close to the treatment site. Each patient was seated in a comfortable position with the affected shoulder exposed, ensuring adequate support and stability throughout the treatment session. Each session lasted approximately 15 minutes.
  Interventions: Other: Therapeutic Exercise Program; Other: Hot Pack; Device: TECAR Therapy; Device: TENS

INTERVENTIONS:
Other: Therapeutic Exercise Program — All patients were administered a therapeutic exercise program that included passive, active-assisted, and active range of motion exercises, stretching, strengthening, and mobilization exercises based on their level of movement restriction and pain intensity for 5 sessions per week for 2 weeks under the supervision of an experienced physiotherapist.
Other: Hot Pack — As part of the treatment protocol, a hot pack was applied to the affected shoulder area for 30 minutes prior to any other therapeutic interventions. This initial application of heat was intended to promote muscle relaxation, increase local blood circulation, and reduce joint stiffness, effectively preparing the shoulder for the subsequent treatments, including therapeutic exercise, TENS and TECAR therapy. The hot pack was maintained at a temperature between 40-45°C, which is considered optimal for achieving therapeutic heat without causing discomfort or skin irritation.
Device: TECAR Therapy — TECAR therapy was administered using the BTL-6000 TR-Therapy PRO device which emitted energy at a frequency of approximately 500 kHz and used three types of electrodes: active, neutral, and static application electrodes. Each patient was seated in a comfortable position with the affected shoulder exposed, ensuring adequate support and stability throughout the treatment session. The affected shoulder was prepared with a conductive gel to enhance energy transfer. During the session, the capacitive electrode was initially applied, targeting the superficial muscles and tendons around the shoulder joint using circular or linear movements for 5 min. Following this, the resistive electrode was employed to target deeper structures, focusing on the joint capsule and rotator cuff muscles for 10 min. The output power was adjusted based on the patient's tolerance, ensuring a comfortable warm sensation without causing discomfort or burning feeling or pain.
  Arms: TECAR combined with TENS and therapeutic exercise and hot pack (TECAR Group)
Device: TENS — TENS was employed as a non-invasive pain management technique in this study, utilizing the Intellect Advanced device manufactured by Chattanooga Group. Electrodes were strategically placed over the affected shoulder, ensuring coverage of the most painful areas as well as relevant nerve pathways to maximize the analgesic effect. A symmetric biphasic waveform was selected, with a frequency of 100 Hz and a pulse duration of 100 microseconds. The intensity of the stimulation was adjusted according to the patient's tolerance, typically aiming for a strong, yet comfortable tingling sensation.

SUMMARY:
Transfer Energy Capacitive and Resistive (TECAR) therapy is a heat therapy method that increases blood circulation at the microscopic level by generating heat in the upper and lower layers of your tissues, reduces inflammation and supports tissue regeneration. In this study, we aimed to evaluate whether this treatment reduces pain and improves functioning in patients with frozen shoulder disease.

DETAILED DESCRIPTION:
Adhesive capsulitis (AC), commonly known as "frozen shoulder," is a prevalent and painful condition resulting from the contracture of the glenohumeral capsule, which significantly impacts individuals' quality of life. While AC is self-limiting in many cases, some patients may experience long-term functional limitations if not treated promptly. One promising intervention is transfer energy capacitive and resistive (TECAR) therapy, which has gained attention for its potential to enhance tissue regeneration, reduce inflammation, and improve pain management by generating heat in superficial and deep tissues. This study aimed to evaluate the effects of TECAR therapy on pain and functional outcomes in patients with adhesive capsulitis (AC).

This prospective, randomized controlled clinical trial included 60 patients [TECAR group: 30, (50.37 ± 13.90 years); control group: 30, (55.27 ± 10.44 years)]. Both groups completed a 2-week tailored therapeutic exercise program, with 30-minute hot pack application and Transcutaneous Electrical Nerve Stimulation. The TECAR group also received three TECAR therapy sessions per week, for a total of six sessions. Pain was measured using the Visual Analog Scale (VAS), functional status with the Shoulder Pain and Disability Index (SPADI), and supraspinatus tendon thickness and bicipital effusion were assessed via ultrasonography. Evaluations were conducted at baseline, 1 and 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were than 18 years of age
* Patients with unilateral shoulder pain of at least 3 on a 10-point Visual Analog Scale (VAS);
* Patients who experienced a more than 50% loss of passive ROM (abduction or external rotation) in the glenohumeral joint relative to the unaffected side
* Patients who had been experiencing the related symptoms for ≥ 3 months.

Exclusion Criteria:

* Patients who had previous shoulder surgery
* Patients who had shoulder injection within the last 3 months
* Patients with inflammatory rheumatic disease,
* Patients with cervical radiculopathy
* Pregnant patients
* Pateints with thyroid disease
* Patients with malignancy,
* Patients who had history of cardiac pacemakers,
* Patients with epilepsy
* Patients who had neurological disease with or without cognitive impairment

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for pain | VAS for pain was applied to the patients before the procedure and at the 4th week and the 12th week after the procedure.
  The Visual Analog Scale (VAS) was employed to evaluate pain intensity in patients. This scale features a 10 cm horizontal line, where one end represents "no pain" (0) and the other represents "worst imaginable pain" (10). Patients were instructed to place a mark on the line that best reflected their current pain level. The distance from the "no pain" end to the patient's mark was measured in centimeters and recorded as the VAS score, providing a numeric representation of their pain intensity

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | SPADI) was applied to the patients before the procedure and at the 4th week and 12th week after the procedure.
  The Shoulder Pain and Disability Index (SPADI) was used to evaluate both pain and functional limitations related to shoulder disorders. SPADI is a patient-reported outcome measure consisting of 13 items, divided into two subscales: pain (5 items) and disability (8 items). Each item is rated on a numerical rating scale (0:no pain or difficulty to 10:worst pain imaginable or extreme difficulty). The scores for each subscale are averaged to create a total score, expressed as a percentage, with higher scores reflecting greater pain and disability. SPADI is widely recognized and validated for assessing shoulder-related pain and functional impairment in both clinical practice and research

OTHER OUTCOMES:
Supraspinatus tendon thickness and bicipital peritendinous effusion | Supraspinatus tendon thickness and bicipital peritendinous effusion were measured using ultrasonography before the study , four weeks after treatment , and 12 weeks later.
  The ultrasonographic assessments were performed using a 5-12 MHz linear array transducer by an expertized physician blinded to the groups. For the Supraspinatus (SS) tendon, the imaging was conducted with the patient in a seated position. To ensure optimal visualization, the patient positioned the hand of the examined side with the palm resting on the ipsilateral hip. The probe was aligned transversely to the inferior aspect of the acromion, allowing both the SS tendon and biceps tendon to appear within the same image. Once the image was captured and frozen, points at 10 mm, 15 mm, and 20 mm lateral to the terminal hyperechoic margin of the biceps tendon were marked. At each marked point, the thickness of the SS tendon was measured. For the biceps tendon, the prob was positioned over the anterior aspect of the shoulder to visualize the bicipital groove and surrounding tissues. This allowed the assessment of peritendinous effusion, with particular attention to any fluid accumulation.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur Uzun, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Physical Medicine and Rehabilitation Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We can share our Study Protocol, Statistical Analysis plan and patients' informed Consent Forms.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will become available starting 6 months after publication.
Access Criteria: The doctors who are specialized in Physical Medicine and Rehabilitation will be able to access upon contact with the principal investigators via email.

REFERENCES:
- [Background] Fields BKK, Skalski MR, Patel DB, White EA, Tomasian A, Gross JS, Matcuk GR Jr. Adhesive capsulitis: review of imaging findings, pathophysiology, clinical presentation, and treatment options. Skeletal Radiol. 2019 Aug;48(8):1171-1184. doi: 10.1007/s00256-018-3139-6. Epub 2019 Jan 3. PMID 30607455
- [Background] Coccetta CA, Sale P, Ferrara PE, Specchia A, Maccauro G, Ferriero G, Ronconi G. Effects of capacitive and resistive electric transfer therapy in patients with knee osteoarthritis: a randomized controlled trial. Int J Rehabil Res. 2019 Jun;42(2):106-111. doi: 10.1097/MRR.0000000000000324. PMID 30362981
- [Background] Paolucci T, Pezzi L, Centra MA, Porreca A, Barbato C, Bellomo RG, Saggini R. Effects of capacitive and resistive electric transfer therapy in patients with painful shoulder impingement syndrome: a comparative study. J Int Med Res. 2020 Feb;48(2):300060519883090. doi: 10.1177/0300060519883090. Epub 2019 Nov 4. PMID 31680597
- [Background] Barassi G, Mariani C, Supplizi M, Prosperi L, Di Simone E, Marinucci C, Pellegrino R, Guglielmi V, Younes A, Di Iorio A. Capacitive and Resistive Electric Transfer Therapy: A Comparison of Operating Methods in Non-specific Chronic Low Back Pain. Adv Exp Med Biol. 2022;1375:39-46. doi: 10.1007/5584_2021_692. PMID 35147930
- [Background] Hawamdeh M. The effectiveness of capacitive resistive diathermy (Tecartherapy®) in acute and chronic musculoskeletal lesions and pathologies. Eur J Sci Res. 2014;118(3):336-40
- [Background] Jain TK, Sharma NK. The effectiveness of physiotherapeutic interventions in treatment of frozen shoulder/adhesive capsulitis: a systematic review. J Back Musculoskelet Rehabil. 2014;27(3):247-73. doi: 10.3233/BMR-130443. PMID 24284277
- [Background] Le HV, Lee SJ, Nazarian A, Rodriguez EK. Adhesive capsulitis of the shoulder: review of pathophysiology and current clinical treatments. Shoulder Elbow. 2017 Apr;9(2):75-84. doi: 10.1177/1758573216676786. Epub 2016 Nov 7. PMID 28405218
- [Background] Vita F, Pederiva D, Tedeschi R, Spinnato P, Origlio F, Faldini C, Miceli M, Stella SM, Galletti S, Cavallo M, Pilla F, Donati D. Adhesive capsulitis: the importance of early diagnosis and treatment. J Ultrasound. 2024 Sep;27(3):579-587. doi: 10.1007/s40477-024-00891-y. Epub 2024 Jun 6. PMID 38844748
- See also: Hawamdeh M. The effectiveness of capacitive resistive diathermy (Tecartherapy®) in acute and chronic musculoskeletal lesions and pathologies. Eur J Sci Res. 2014;118(3):336-40 — https://www.semanticscholar.org/paper/The-effectiveness-of-Capacitive-Resistive-Diathermy-Hawamdeh/b5d02c41a382e1d9043d3d4f6ed9f2f5e9797737